CLINICAL TRIAL: NCT05633979
Title: Phase 1b Study of EZH1/2 Inhibitor Valemetostat in Combination With Trastuzumab Deruxtecan in Subjects With HER2 Low/Ultra-low/Null Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0315; NCI-2022-09968 (Other: NCI-CTRP Clinical Trial Registry)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will receive the same drugs at the same schedule, and the same dose of trastuzumab deruxtecan
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Valemetostat
- Group 2 (Experimental): Participants will only receive 1 dose level of valemetostat.
  Interventions: Drug: Valemetostat

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Given by IV (vein)
  Arms: Group 1
Drug: Valemetostat — Given by PO

SUMMARY:
To find a recommended dose of valemetostat that can be given in combination with trastuzumab deruxtecan to patients with low/ultra-low HER2-expressing metastatic breast cancer.

DETAILED DESCRIPTION:
Primary Objectives:

Dose escalation part:

1. To evaluate the safety and determine the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) of valemetostat in combination with trastuzumab deruxtecan (T-DXd).

   Dose expansion part:
2. To evaluate the objective response rate (ORR) of valemetostat at the RDE in combination with T-DXd.

Secondary Objectives:

Dose escalation:

1. To determine ORR; defined as a percentage of subjects who achieve complete response (CR) or partial response (PR) by RECIST 1.1 criteria.
2. To determine survival outcomes, including duration of response (DoR), progression free survival (PFS), and overall survival (OS).
3. To determine the Clinical Benefit Rate (CBR) defined as stable disease (SD) ≥ 16 weeks + PR + CR.

Dose expansion:

1. To determine survival outcomes, including DoR, PFS, and OS.

   * DOR of the proposed treatment: the time from observing response to the valemetostat treatment until objective tumor progression (PD)
   * PFS: the time from starting valemetostat treatment until objective tumor progression (PD) or death due to any cause.
   * Overall survival (OS): the time from starting valemetostat treatment until death due to any cause.
2. To determine the CBR defined as SD ≥16 weeks + PR + CR.
3. To evaluate safety of valemetostat in combination with T-DXd.
4. To evaluate the pharmacokinetics (PK) of both the drugs in combination.
5. To evaluate the immunogenicity of T-DXd

Exploratory Objectives:

1. To investigate pharmacodynamic biomarkers.
2. To investigate biomarkers that may aid in identifying subjects who may derive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age or the minimum legal adult age (whichever is greater) at the time the informed consent form (ICF) is signed.
2. Pathologically confirmed HER2 low/ultra-low/null breast cancer. HER2 low is defined as IHC 2+/ISH- or IHC 1+/(ISH- or undefined), HER2 ultra-low is defined as IHC 0 with detectable faint/barely perceptible incomplete staining in ≤10% tumor cells and HER2 null is defined as IHC 0 without any observed tumor cell staining, regardless of hormone receptor expression status, and as determined by the Ventana 4B5 IHC assay The accrual numbers of HER2 ultra-low/null and HER2 low should be approximately 1:1 in the dose-escalation and dose-expansion cohort (i.e., 6 subjects for HER2 ultra-low/null and 6 subjects for HER2 low in dose-escalation cohort, 10 subjects for HER2 ultra-low/null and 10 subjects for HER2 low in dose-expansion cohort). Initial subject inclusion may be based on previously obtained HER2 testing results, however final HER2 status determination (HER2 low, ultra-low, or null) will be based on centralized pathologist (re)evaluation of HER2 IHC staining using the Ventana 4B5 assay at MDA Department of Pathology laboratory.

   If HER2 eligibility assessment and subject inclusion are based on results from a previous HER2 IHC test performed with an IHC assay different from the Ventana 4B5 assay, or if the IHC slides from the initial test are not available for re-evaluation, adequate material for HER2 testing using the Ventana 4B5 assay must be provided to MDA Department of Pathology laboratory.
3. MBC or locally progressive breast cancer that is not a surgical candidate.
4. Has progressed on and would no longer benefit from endocrine therapy in hormone receptor-positive subjects.
5. Has been treated with at least 1 prior line of chemotherapy in the metastatic or locally progressive setting.
6. Has adequate treatment washout period by the time of enrollment, defined as:

   Treatment Washout Period Major surgery ≥ 4 weeks Radiation therapy including palliative stereotactic radiation to chest ≥ 4 weeks Palliative stereotactic radiation therapy to other anatomic areas ≥ 2 weeks Anti-cancer chemotherapy (Immunotherapy [non-antibody based therapy]), retinoid therapy, hormonal therapy
   * 3 weeks Targeted agents and small molecules ≥ 2 weeks or 5 half-lives, whichever is longer Nitrosoureas or mitomycin C ≥ 6 weeks Antibody-based anti-cancer therapy ≥ 4 weeks Chloroquine/Hydroxychloroquine >14 days
7. Has at least one measurable lesion per RECIST (except for up to the first 5 subjects who enroll in dose escalation part where the measurable lesions meeting RECIST definition are not mandatory).
8. Is willing to provide fresh tumor tissue via tumor biopsy only if the participant has a disease that can be safely accessed through a CT-guided/US-guided or percutaneous biopsy for multiple core biopsies judged by the investigator. If the participant doesn't have a disease that can be safely accessed, they are still eligible.
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
10. Negative serum pregnancy test within 72 hours of receiving the first dose of the study medication for women of childbearing potential as per institutional guidelines. Post-menopausal women (defined as having no menses for at least 1 year) and surgically sterilized women are not required to undergo pregnancy tests.
11. Subjects of childbearing potential must be willing to use effective birth control methods or be surgically sterile or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of the study drug (for males) and 7 months after last dose of study drug (for females). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for at least 1 year.
12. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 3 months after the final study drug administration.
13. Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and for at least 3 months after the final study drug administration.
14. The patient must have adequate organ function as determined by the following laboratory values:

    1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × the upper limit of normal (ULN). For those with liver metastasis, ALT and AST ≤5.0 × ULN.
    2. Total bilirubin ≤1.5 × ULN, except for subjects with Gilbert's syndrome (e.g., a gene mutation in UGT1A1), who can have total bilirubin <3.0 mg/dL.
    3. Absolute neutrophil count (ANC) ≥1500/mm3 (granulocyte colony-stimulating factor administration is not allowed within 1 week prior to Screening assessment).
    4. Hemoglobin ≥9.0 g/dL (red blood cell transfusion is not allowed within 1 week prior to Screening assessment).
    5. Platelet count ≥100,000/mm3 (Platelet transfusion is not allowed within 1 week prior to Screening assessment).
    6. Creatinine clearance ≥30 mL/min (measured by the Cockcroft-Gault equation*).

       * Female: ([140-age] × weight in kg)/(serum creatinine × 72) × 0.85 Male: ([140-age] × weight in kg)/(serum creatinine × 72)
    7. Serum Albumin ≥ 2.5 g/dL
15. Acute non-hematologic toxic effects (as evaluated by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 5.0) of any prior therapy (except alopecia) resolved as shown below:

    1. Peripheral neuropathy: Grade ≤2
    2. Fatigue: Grade ≤2
    3. All others: Grade ≤1

Exclusion Criteria:

1. Has previously been treated with any anti-HER2 therapy, including T-DXd, or EZH inhibitors.
2. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study registration.
3. Prior malignancy active within the previous 2 years except for locally curable cancer that is currently considered as cured, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer
4. Uncontrolled or significant cardiovascular disease, including the following:

   1. LVEF < 50% within 28 days
   2. Evidence of prolongation of QT/QTc (e.g., repeated episodes of QT corrected for heart rate using Fridericia's method [QTcF] >450 ms) (average of triplicate determinations; over a 5 min time window when the subject has been supine position for at least 10 min without any environmental stimuli).
   3. Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome
   4. History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
   5. Uncontrolled arrhythmia (subjects with asymptomatic, controllable atrial fibrillation may be enrolled), or asymptomatic persistent ventricular tachycardia
   6. Subject has clinically relevant bradycardia of 50 bpm unless the subject has a pacemaker
   7. History of second or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers, within 6 months prior to Screening
   8. Myocardial infarction within 6 months prior to Screening
   9. Angioplasty or stent graft implantation within 6 months prior to Screening
   10. Uncontrolled angina pectoris within 6 months prior to Screening
   11. New York Heart Association (NYHA) Class 2-4 congestive heart failure
   12. Coronary/peripheral artery bypass graft within 6 months prior to Screening
   13. Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg)
   14. Complete left or right bundle branch block
5. Systemic treatment with corticosteroids (>10 mg daily prednisone equivalents). Note: Short-course systemic corticosteroids (e.g., prevention/treatment for transfusion reaction) or use for a non-cancer indication (e.g., adrenal replacement) is permissible.
6. Female who is pregnant or breastfeeding or intends to become pregnant during the study
7. Has known human immunodeficiency virus (HIV) infection or active hepatitis B or C infection (screen test is not required). Subjects positive for hepatitis C (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.
8. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection requiring treatment with intravenous antibiotics, antivirals, or antifungals. Note: Subjects with localized fungal infections of skin or nails are eligible.
9. Any active uncontrolled systemic diseases or other medical conditions considered to be poorly controlled by the investigator, including, but not limited to, bleeding diatheses
10. A history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
11. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study registration, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.).
12. Any autoimmune, connective tissue or inflammatory disorders (e.g., rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for subjects who are included in the study.
13. Current use of moderate or strong cytochrome P450 (CYP)3A inducers (Table 17)
14. Prior complete pneumonectomy
15. Medical history or complication considered inappropriate for participation in the study, or a serious physical or psychiatric disease, the risk of which may be increased by participation in the study in the investigator's opinion
16. A history of substance abuse or medical conditions such as clinically significant cardiac or pulmonary diseases or psychological conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
17. Known or suspected hypersensitivity to valemetostat and T-DXd or any of the excipients.
18. Subjects with symptomatic brain metastases, or subjects with treated brain metastases that are no longer symptomatic but who require treatment with steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
The Overall Response Rate (ORR) | through study completion; an average of 2-3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Damodaran, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://WWW.mdanderson.org